CLINICAL TRIAL: NCT01643330
Title: A Phase 2b, Double-Blind, Placebo-Controlled, Multinational, Multicenter, Randomized Study Evaluating the Safety and Efficacy of Intracoronary Administration of MYDICAR® (AAV1/SERCA2a) in Subjects With Heart Failure
Brief Title: A Study of Genetically Targeted Enzyme Replacement Therapy for Advanced Heart Failure
Acronym: CUPID-2b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celladon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELL-004; 2012-001700-37 (EudraCT Number)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Ischemic Cardiomyopathy; Non-ischemic Cardiomyopathy; Heart Failure; Cardiomyopathies
Keywords: Cardiomegaly; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Cardiomegaly; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AAV1/SERCA2a (MYDICAR) (Experimental): Intracoronary infusion
  Interventions: Genetic: AAV1/SERCA2a (MYDICAR)
- Placebo (Placebo Comparator): Intracoronary infusion
  Interventions: Genetic: Placebo

INTERVENTIONS:
Genetic: AAV1/SERCA2a (MYDICAR) — Single intracoronary infusion 1 x 10^13 DNase Resistant Particles (DRP) MYDICAR
  Arms: AAV1/SERCA2a (MYDICAR)
Genetic: Placebo — Single intracoronary infusion
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess whether MYDICAR can reduce the frequency and/or delay heart failure related hospitalizations in persons with advanced heart failure when added to their maximal and optimized therapy.

ELIGIBILITY:
Inclusion Criteria:

Unless otherwise specified, screening must be performed within 30 days prior to administration of investigational medicinal product on Day 0 except as noted under Inclusion Criteria #1 and 4. Subjects must meet the following criteria to be eligible for the study:

1. Negative neutralizing AAV1 antibodies (NAb) (titer <1:2 or equivocal) within 90 days of screening.
2. 18-80 years of age, inclusive, at the time of signing the informed consent.
3. Chronic systolic HF due to ischemic or non-ischemic cardiomyopathy. Subjects with ischemic cardiomyopathy must have at least one major coronary vessel with Thrombolysis in Myocardial Infarction (TIMI) grade 3 flow. If a subject has not undergone coronary angiography within 2 months, this criterion may be assessed after the subject is randomized and undergoes angiography just prior to the planned infusion of investigational medicinal product.

   1. Hypertrophic cardiomyopathy is excluded.
   2. Toxic and alcoholic cardiomyopathies are allowed as long as toxin or alcohol exposure has been eliminated and a sufficient amount of limit has elapsed to rule-out spontaneous recovery.
4. Left ventricular ejection fraction (LVEF) ≤35% anytime during the 60-day window prior to administration of investigational medicinal product.
5. Diagnosis of New York Heart Association (NYHA) class II, III or IV HF for a minimum of 90 days prior to screening.
6. Individualized, maximal, optimized HF therapy consistent with American College of Cardiology (ACC)/American Heart Association (AHA) and European Society of Cardiology (ESC) practice guidelines for the treatment of chronic heart failure (ACC/AHA/ESC HF guidelines) and as updated from time to time:

   1. Medical therapy as appropriate to the individual subject including oral diuretic, angiotensin-converting enzyme (ACE) inhibitor (or angiotensin-receptor blocker (ARB) if ACE intolerant) and, as tolerated, beta blocker at approved dosages as labeled in the respective package insert. The choice of beta blocker is limited to those approved for heart failure in all participating countries (bisoprolol, carvedilol or sustained release metoprolol succinate). Unless contraindicated or not tolerated, the addition of an aldosterone antagonist should be considered in the absence of hyperkalemia and significant renal dysfunction and according to evolving standards; the final decision is at the discretion of the investigator. Dosing of the above medications must be stable for a minimum of 30 days prior to screening, although up- or down-titration of diuretics, as medically indicated, is permitted. Enrollment of any subject with any deviation from this combination must be preapproved by the medical monitor.
   2. Resynchronization therapy, if clinically indicated according to ACC/AHA/ESC HF guidelines, must have been implanted at least 6 months prior to screening.
   3. Implantable cardioverter defibrillator (ICD), if clinically indicated according to ACC/AHA/ESC HF guidelines, must have been implanted a minimum of 30 days prior to screening.
   4. Cardiac rehabilitation should be consistent with the Agency for Health Care Policy and Research Clinical Practice Guideline, Number 17, Cardiac Rehabilitation. This does not imply that the potential candidate must be enrolled in a cardiac rehabilitation program at screening or in the future.
7. All women of childbearing potential must have a negative urine pregnancy test prior to administration of investigational medicinal product and agree to use adequate contraception (defined as oral or injectable contraceptives, intrauterine devices, surgical sterilization or a combination of a condom and spermicide) or limit sexual activity to vasectomized partner for 3 months after administration of investigational medicinal product. Men capable of fathering a child must agree to use barrier contraception (combination of a condom and spermicide) or limit activity to post-menopausal, surgically sterilized, or a contraception-practicing partner, for 3 months after administration of investigational medicinal product.
8. Ability to understand and comply with study requirements as evidenced by providing signed written informed consent form and Release of Medical Information Form.
9. Presence of at least one of the following risk factors:

   1. Hospitalization for heart failure within 6 months of screening, or in lieu of hospitalization, at least 2 outpatient interventions for the intended treatment of signs and symptoms of worsening heart failure (e.g., intravenous diuretics, peripheral ultrafiltration)
   2. N-terminal pro-B-type natriuretic peptide (NT-proBNP) >1200 pg/mL (BNP >225 pg/mL) within 30 days of screening; if subject is in atrial fibrillation, NT-proBNP >1600 pg/mL (BNP >275 pg/mL) within 30 days of screening
10. In Germany only: Medically indicated for diagnostic angiography at the clinician's discretion.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Any intravenous (IV) therapy with positive inotropes, vasodilators or diuretics within 30 days prior to screening.
2. Restrictive cardiomyopathy, obstructive cardiomyopathy, acute myocarditis, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease or discrete LV aneurysm.
3. Cardiac surgery, percutaneous coronary intervention (PCI) or valvuloplasty within 30 days prior to screening.
4. Myocardial infarction (MI) (e.g., ST elevation MI [STEMI] or large non-STEMI) within 90 days prior to screening. Large non-STEMI shall be defined >3x upper limit of normal (ULN) for creatinine kinase (CK)-MB or >5x ULN for troponin.
5. Prior heart transplantation, left ventricular reduction surgery (LVRS), cardiomyoplasty, passive restraint device (e.g., CorCap™ Cardiac Support Device), surgically implanted left ventricular assist device (LVAD) or cardiac shunt.
6. Likely need for an immediate heart transplant or LVAD implant due to hemodynamic instability.
7. Prior coronary artery bypass grafting (CABG) is not considered ideal for inclusion in the study; however, a potential candidate can be reviewed on a case-by-case basis. Ideally, the orifice of the graft should be easy to engage with a catheter and the graft should perfuse a significant amount of potentially viable myocardium.
8. Known hypersensitivity to contrast agents used for angiography; history of, or likely need for, high dose steroid pretreatment prior to contrast angiography.
9. Significant, in the opinion of the investigator, left main or ostial right coronary luminal stenosis.
10. Liver function tests (alanine amino transferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase) >3x ULN within 30 days prior to investigational medicinal product administration or known intrinsic liver disease (e.g., cirrhosis, chronic hepatitis B or hepatitis C virus infection).
11. Current or likely need for hemodialysis within 12 months following enrollment or current glomerular filtration rate (GFR) ≤20 mL/minute/1.73 m^2 estimated by Modification of Diet in Renal Disease (MDRD) calculation.
12. Bleeding diathesis or thrombocytopenia defined as platelet count <50,000 platelets/μL.
13. Anemia defined as hemoglobin <9 g/dL, provided that there is no evidence of bleeding.
14. Known AIDS or HIV seropositive status, or a previous diagnosis of immunodeficiency with an absolute neutrophil count <1000 cells/mm^3.
15. Diagnosis of, or treatment for, any cancer other than basal cell carcinoma within the last 5 years. (Past medical history of cancer is not exclusionary as long as subject has been disease-free for at least 5 years since the time of diagnosis and treatment).
16. Previous participation in a study of gene transfer; however, if the study was unblinded or documentation otherwise exists that the subject was randomized to the placebo control group and did not receive active gene transfer agent, the subject may be considered for this study.
17. Receiving investigational intervention or participating in another clinical study within 30 days or within 5 half-lives of the investigational drug administration prior to screening. Exception may be made if the individual is enrolled in a non-therapeutic observational study (registry) or the observational portion of a therapeutic study where the sponsoring authority authorizes enrollment.
18. Pregnant or breast-feeding.
19. Recent history of psychiatric disease, including drug or alcohol abuse, that is likely to impair, in the opinion of the investigator, the subject's ability to comply with protocol-mandated procedures.
20. Other concurrent medical condition(s) that, while not explicitly excluded by the protocol, could jeopardize the safety of the subject or objectives of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Time to recurrent events (heart failure [HF]-related hospitalizations, ambulatory worsening HF) in the presence of terminal events (all-cause death, heart transplant, mechanical circulatory support device [MCSD] implantation) | From administration up to 12 months

SECONDARY OUTCOMES:
Time-to-terminal event (all-cause death, heart transplant, MCSD implantation) in the presence of recurrent events. | From administration up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-858-366-4288, Study Director — Celladon Corporation
Locations (54):
- United States (29):
  - Birmingham, Alabama
  - La Jolla, California
  - Long Beach, California
  - San Diego, California
  - Sylmar, California
  - Newark, Delaware
  - Jacksonville, Florida
  - Miami, Florida
  - Augusta, Georgia
  - Iowa City, Iowa
  - Alexandria, Louisiana
  - Boston, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - New York, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Rapid City, South Dakota
  - Germantown, Tennessee
  - Tullahoma, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Tacoma, Washington
  - Waukesha, Wisconsin
- Belgium (2):
  - Aalst
  - Leuven
- Denmark (3):
  - Aalborg
  - Coppenhagen
  - Hvidovre
- Germany (5):
  - Bad Nauheim
  - Berlin
  - Cologne
  - Dresden
  - München
- Hungary (2):
  - Budapest
  - Debrecen
- Israel (4):
  - Ashkelon
  - Holon
  - Jerusalem
  - Rehovot
- Groningen, Netherlands
- Poland (3):
  - Gdansk
  - Wroclaw
  - Zabrze
- Sweden (3):
  - Malmo
  - Örebrö
  - Stockholm
- United Kingdom (2):
  - Glasgow
  - London

REFERENCES:
- [Background] Jaski BE, Jessup ML, Mancini DM, Cappola TP, Pauly DF, Greenberg B, Borow K, Dittrich H, Zsebo KM, Hajjar RJ; Calcium Up-Regulation by Percutaneous Administration of Gene Therapy In Cardiac Disease (CUPID) Trial Investigators. Calcium upregulation by percutaneous administration of gene therapy in cardiac disease (CUPID Trial), a first-in-human phase 1/2 clinical trial. J Card Fail. 2009 Apr;15(3):171-81. doi: 10.1016/j.cardfail.2009.01.013. PMID 19327618
- [Background] Jessup M, Greenberg B, Mancini D, Cappola T, Pauly DF, Jaski B, Yaroshinsky A, Zsebo KM, Dittrich H, Hajjar RJ; Calcium Upregulation by Percutaneous Administration of Gene Therapy in Cardiac Disease (CUPID) Investigators. Calcium Upregulation by Percutaneous Administration of Gene Therapy in Cardiac Disease (CUPID): a phase 2 trial of intracoronary gene therapy of sarcoplasmic reticulum Ca2+-ATPase in patients with advanced heart failure. Circulation. 2011 Jul 19;124(3):304-13. doi: 10.1161/CIRCULATIONAHA.111.022889. Epub 2011 Jun 27. PMID 21709064
- [Background] Horowitz JD, Rosenson RS, McMurray JJ, Marx N, Remme WJ. Clinical Trials Update AHA Congress 2010. Cardiovasc Drugs Ther. 2011 Feb;25(1):69-76. doi: 10.1007/s10557-011-6285-9. PMID 21340529
- [Background] Zsebo K, Yaroshinsky A, Rudy JJ, Wagner K, Greenberg B, Jessup M, Hajjar RJ. Long-term effects of AAV1/SERCA2a gene transfer in patients with severe heart failure: analysis of recurrent cardiovascular events and mortality. Circ Res. 2014 Jan 3;114(1):101-8. doi: 10.1161/CIRCRESAHA.113.302421. Epub 2013 Sep 24. PMID 24065463
- [Background] Greenberg B, Butler J, Felker GM, Ponikowski P, Voors AA, Pogoda JM, Provost R, Guerrero J, Hajjar RJ, Zsebo KM. Prevalence of AAV1 neutralizing antibodies and consequences for a clinical trial of gene transfer for advanced heart failure. Gene Ther. 2016 Mar;23(3):313-9. doi: 10.1038/gt.2015.109. Epub 2015 Dec 24. PMID 26699914
- [Result] Greenberg B, Butler J, Felker GM, Ponikowski P, Voors AA, Desai AS, Barnard D, Bouchard A, Jaski B, Lyon AR, Pogoda JM, Rudy JJ, Zsebo KM. Calcium upregulation by percutaneous administration of gene therapy in patients with cardiac disease (CUPID 2): a randomised, multinational, double-blind, placebo-controlled, phase 2b trial. Lancet. 2016 Mar 19;387(10024):1178-86. doi: 10.1016/S0140-6736(16)00082-9. Epub 2016 Jan 21. PMID 26803443
- [Derived] Greenberg B, Yaroshinsky A, Zsebo KM, Butler J, Felker GM, Voors AA, Rudy JJ, Wagner K, Hajjar RJ. Design of a phase 2b trial of intracoronary administration of AAV1/SERCA2a in patients with advanced heart failure: the CUPID 2 trial (calcium up-regulation by percutaneous administration of gene therapy in cardiac disease phase 2b). JACC Heart Fail. 2014 Feb;2(1):84-92. doi: 10.1016/j.jchf.2013.09.008. Epub 2014 Jan 25. PMID 24622121